CLINICAL TRIAL: NCT02365415
Title: Systemic Rapamycin (Sirolimus) to Prevent In-Stent Restenosis Following Pulmonary Artery Stent Placement
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll appropriate patients
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jesse J Esch, Staff Cardiologist, Instructor in Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00005257
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Pulmonary Stenosis; In-stent Stenosis
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus (Experimental): Patients randomized to this arm will receive 8 weeks of enteral Rapamycin (sirolimus), with dosage titrated to achieve target blood levels.
  Interventions: Drug: Sirolimus
- Control (No Intervention): No treatment.

INTERVENTIONS:
Drug: Sirolimus — 8 weeks oral sirolimus, following drug levels
  Other Names: Rapamycin, Rapamune
  Arms: Sirolimus

SUMMARY:
This is a research study to assess whether an oral medication can benefit some patients being treated for peripheral pulmonary stenosis (PPS), which is narrowing of the blood vessels that send blood to the lungs (pulmonary arteries).

In the cardiac catheterization laboratory, the investigators treat PPS by dilating the narrowed segments of pulmonary arteries using balloon catheters. Sometimes the investigators also place stents which are mesh tubes that help keep the narrowed vessel open. Some stents suffer from in-growth of tissue into the stents which causes recurrent obstructions inside the stent (i.e. making the opening inside the mesh tube narrow again), so called in-stent stenosis (ISS).

The purpose of this study is to use a medication that is approved for use in children (for a different purpose) to decrease the amount of cell ingrowth inside the stents (i.e. decrease the problematic in-stent stenosis). The medication is called rapamycin, also known as sirolimus (trade name Rapamune). It has antiproliferative properties which means that it slows down cell division which the investigators believe cause the recurrent narrowing inside stents.

Rapamycin is a medicine that can be taken by mouth as a liquid or pill or via a feeding tube. There will still be a need for interventions in the catheterization laboratory but the investigators hope that by taking this medicine some children would need fewer catheterizations in the future. Our early experiences with a few patients who have been treated with rapamycin due to in-stent stenosis in the pulmonary arteries suggest that it may be helpful.

In this study, patients and families who are interested in possibly trying this new approach will be randomized to sirolimus or no sirolimus. The investigators will compare the developement of ISS over time between these groups, in a hope to learn whether oral sirolimus reduces ISS development.

DETAILED DESCRIPTION:
This is a research study to assess whether an oral medication can benefit some patients being treated for peripheral pulmonary stenosis (PPS). PPS, which can be associated with several different congenital heart diseases, is narrowing of the blood vessels that send blood to the lungs (pulmonary arteries) to pick up oxygen before returning the blood to the heart and the rest of the body. The right ventricle (RV) is the pumping chamber that pumps blood into the pulmonary arteries and the lungs.

PPS can result in high RV pressure, reduced blood flow to one lung, or uneven blood flow within either lung. If left untreated these abnormalities place affected children at risk for abnormal RV function and failure of this pumping chamber which may be seen as decreased ability to do exercise, heart rhythm problems, fainting, or even death.

In the cardiac catheterization laboratory, the investigators treat PPS by dilating the narrowed segments of pulmonary arteries using balloon catheters. Sometimes the investigators also place stents which are mesh tubes that help keep the narrowed vessel open. Some stents suffer from in-growth of tissue into the stents which causes recurrent obstructions inside the stent (i.e. making the opening inside the mesh tube narrow again), so called in-stent stenosis (ISS). This effectively causes recurrent PPS and recurrence of the associated risks listed above.

The purpose of this study is to use a medication that is approved for use in children (for a different purpose) to decrease the amount of cell ingrowth inside the stents (i.e. decrease the problematic in-stent stenosis). The medication is called rapamycin, also known as sirolimus (trade name Rapamune), and has been used safely for many years in children and adults after organ transplantation to prevent rejection of the new organ. It has antiproliferative properties which means that it slows down cell division which the investigators believe cause the recurrent narrowing inside stents. By slowing down the cell division the investigators believe that the stents will stay open instead of becoming narrowed inside again. This medicine is found in many types of stents placed in adults with narrowed arteries around the heart (so called drug-eluding stents) and appear to help keep these blood vessels open after heart attacks (or to prevent heart attacks). Such stents are currently not available for pulmonary arteries; therefore the investigators give the medicine by mouth instead (which has also been used in adults with stents in narrowed arteries around the heart).

Rapamycin is a medicine that can be taken by mouth as a liquid or pill or via a feeding tube. There will still be a need for interventions in the catheterization laboratory but the investigators hope that by taking this medicine some children would need fewer catheterizations in the future. The investigators believe it may help lessen the risk of recurrent in-stent stenosis and the associated problems listed above. Our early experiences with a few patients at BCH who have been treated with rapamycin due to in-stent stenosis in the pulmonary arteries suggest that it may be helpful.

In this study, patients and families who are interested in possibly trying this new approach will be randomized to sirolimus or no sirolimus. The investigators will compare the developement of ISS over time between these groups, in a hope to learn whether oral sirolimus reduces ISS development.

ELIGIBILITY:
Inclusion Criteria:

* In-stent stenosis: At least one stent from at least one prior catheterization affected by in-stent stenosis (≥25% stenosis and a diameter narrower or equal to the distal vessel).
* At least one of the following:

  * RV hypertension: At least one half systemic RVp or ≥ 70 mm Hg by echocardiogram or per baseline hemodynamics on most recent catheterization
  * Pulmonary blood flow maldistribution: ≤ 25% of flow to either lung or regional decrease in individual lobar segments.
  * Pulmonary hypertension: Mean PA pressure ≥ 20 mmHg in unobstructed segments by most recent catheterization.
* Informed consent of patient and/or parent/guardian
* Agreement to participate in protocol, including follow-up testing

Exclusion Criteria:

* Age ≤ 6 months
* Pulmonary artery surgery or transcatheter PA dilations in the past 6 weeks.
* Malignancy (past or present)
* Active infection
* Pregnancy (current or planned within the next 1 year)
* Organ dysfunction as evidenced by laboratory abnormalities

  * Renal: BUN > 40 mg/dL, or Cr > normal limit for age (by powerchart). Exceptions can be made at the discretion of the study physician if BUN or Cr elevation is known to be due to diuretic management with plan to reduce dosing, or other reversible mechanism.
  * Hepatic: AST or ALT > 120 unit/L, or total bilirubin > 3 mg/dL
  * Immune: WBC < 2,000, or ANC or ALC < 1,000
  * Hematologic: Hgb< 7 g/dL, or Hct< 21%, or platelet count < 80,000. Exceptions can be made at the discretion of the study physician if plans include transfusion of blood products in the catheterization laboratory and a known reversible etiology for the anemia.
* Lipids: Total cholesterol > 250 mg/dL, HDL < 30 g/dL

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Percent change in in-stent stenosis | 6 months

SECONDARY OUTCOMES:
RV pressure | 6 months
Adverse drug event | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Marshall, MD, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No